CLINICAL TRIAL: NCT06639958
Title: Risk-Based 6MP Adherence Enhancement Strategies in Children, Adolescent and Young Adults With ALL - A Pilot Study
Brief Title: A Study of Different Programs to Help ALL Patients With Taking Maintenance Medicine at Home
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: All potential pilot phase pts have been enrolled.
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ACCL2433; NCI-2024-08458 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCL2433 (Other: Children's Oncology Group); COG-ACCL2433 (Other: DCP); ACCL2433 (Other: CTEP); UG1CA189955 (NIH)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia; Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Specimen Handling; Health Promotion; Educational Status; Mercaptopurine; azathiopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adherers arm III (EDU) (Experimental): Patients receive another Patient Supply Kit and MEMS® TrackCap™ to use on day 1 of Maintenance cycle 3 and for the remaining duration of the study. Patients and their caregiver view the MIPE program that features video clips of ALL patients and their parents/other adults discussing Maintenance treatment in the clinic on day 1 of cycle 3. Additionally, patients undergo blood sample collection on the study.
  Interventions: Procedure: Biospecimen Collection; Other: Informational Intervention; Other: Media Intervention; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Behavioral: Training and Education
- Adherers arm IV (pIP) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Behavioral: Compliance Monitoring; Other: Informational Intervention; Other: Media Intervention; Other: Medical Device Usage and Evaluation; Drug: Mercaptopurine; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention; Behavioral: Training and Education
- Non-adherers arm I (IP) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Behavioral: Compliance Monitoring; Other: Health Promotion and Education; Other: Informational Intervention; Other: Media Intervention; Other: Medical Device Usage and Evaluation; Drug: Mercaptopurine; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention; Behavioral: Training and Education
- Non-adherers arm II (U-iIP) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Behavioral: Compliance Monitoring; Other: Health Promotion and Education; Other: Informational Intervention; Other: Media Intervention; Other: Medical Device Usage and Evaluation; Drug: Mercaptopurine; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention; Behavioral: Training and Education

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Behavioral: Compliance Monitoring — Receive DST
  Arms: Adherers arm IV (pIP); Non-adherers arm I (IP)
Behavioral: Compliance Monitoring — Healthcare provider reviews DST response rates with the patient and any challenges they are having with 6MP adherence every 4 weeks at clinic visits
  Arms: Non-adherers arm II (U-iIP)
Other: Health Promotion and Education — Receive customized printed medication schedules
  Arms: Non-adherers arm I (IP); Non-adherers arm II (U-iIP)
Other: Informational Intervention — Receive Patient Supply Kit
Other: Media Intervention — View MIPE program videos
Other: Media Intervention — Review booster MIPE videos
  Arms: Non-adherers arm II (U-iIP)
Other: Medical Device Usage and Evaluation — Use MEMS® with TrackCap™
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
  Arms: Adherers arm IV (pIP); Non-adherers arm I (IP); Non-adherers arm II (U-iIP)
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive automated customized electronic reminders via smartphone
  Arms: Non-adherers arm I (IP); Non-adherers arm II (U-iIP)
Behavioral: Telephone-Based Intervention — Receive additional automated reminders
  Arms: Non-adherers arm II (U-iIP)
Behavioral: Telephone-Based Intervention — Manually activate daily smartphone reminders with successive alerts (using the "snooze" function)
  Arms: Adherers arm IV (pIP)
Behavioral: Telephone-Based Intervention — Receive electronic reminders with successive alerts (using the "snooze" function)
  Arms: Adherers arm IV (pIP)
Behavioral: Training and Education — Undergo training for prompting and supervising 6MP

SUMMARY:
This clinical trial tests different programs to help patients with acute lymphoblastic leukemia (ALL) remember to take their medications during maintenance therapy at home. One problem with ALL maintenance treatment is remembering to take medicines at home like patients are supposed to. In maintenance, a medicine called 6-mercaptopurine or "6MP" is taken by mouth every day at home. In this study, 6MP prescriptions are filled into a special medication bottle called MEMS® which is fitted with a special cap called TrackCap™ that electronically records when the medication bottle is opened. Researchers are trying a new program to help patients be better at taking their 6MP like they're supposed to. This new program may help patients to remember to take their 6MP medication.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Collect data on the feasibility of a phase 3 adherence-enhancing 2 parallel 2-arm randomized clinical trial.

Ia. Estimate participation rates, refusal reasons, and attrition rates. Ib. Evaluate rates of completeness of all aspects of the study (surveys [rates of missing elements]; MEMS® TrackCap™ return rates; maintenance form return rates from site clinical research assistants [CRAs]; blood samples for pharmacogenetics and deoxyribonucleic acid [DNA]-incorporated thioguanine nucleotide [DNA-TG] levels).

SECONDARY OBJECTIVES:

I. Among baseline non-adherers, estimate the impact of ultra-intensified intervention package (U-iIP) versus (vs.) intervention package (IP) on 6MP adherence.

II. Among baseline adherers, estimate the impact of patient-empowered intervention package (pIP) vs. education alone (EDU) on 6MP adherence.

OUTLINE:

Patients receive the Patient Supply Kit containing an empty MEMS® medication bottle with TrackCap™ with child resistant medication bottles and child resistant standard caps, and written instructions for the patient and pharmacist, along with their 6MP prescription. Beginning on day 1 cycle 1 of Maintenance Therapy, patients start using the MEMS® medication bottle with TrackCap™. Clinical research assistants contact patients and parents by telephone the next day to confirm that TrackCap™ is being used, to identify any obstacles, and to determine solutions. Patients are instructed to return the first MEMS® TrackCap™ to the clinic on day 1 of Maintenance cycle 2. Patients are then assigned to 1 of 2 groups based on baseline adherence rates (adherers [adherence rate >= 95%] and non-adherers [adherence rate < 95%]).

NON-ADHERERS: Patients are randomized to 1 of 2 arms during cycle 2 of Maintenance therapy.

ARM I (IP): Patients receive another Patient Supply Kit and MEMS® TrackCap™ to use on day 1 of Maintenance cycle 3 and for the remaining duration of the study. Patients and their caregiver view the multimedia interactive patient/parent/other adult education (MIPE) program that features video clips of ALL patients and their parents/other adults discussing Maintenance treatment in the clinic on day 1 of cycle 3. A designated parent/other adult is selected and trained briefly in prompting and supervising the patient to take 6MP daily by the CRA on day 1 of Maintenance cycle 3. Patients also receive customized printed medication schedules approximately every 4 weeks (days 1, 29, and 57) during Maintenance cycles 3-5 (during scheduled clinic visits) from their healthcare provider. Patients and/or the parent/other adult receive automated customized electronic reminders delivered via smartphone according to the patient's electronic 6MP schedule. Once the designated parent/other adult receives the customized electronic reminder for 6MP, they are instructed to prompt initiation of the 6MP dose (if necessary), and to supervise the ingestion of the prescribed 6MP (in all instances). If the patient is not present when the dose of 6MP is due, the patient receives a call from the designated parent/other adult to prompt initiation of the dose. Patients and designated parents/other adults will be instructed to electronically indicate when 6MP has been taken (indicative of directly supervised therapy [DST] execution). Additionally, patients undergo blood sample collection on the study.

ARM II (U-iIP): Patients receive another Patient Supply Kit and MEMS® TrackCap™ to use on day 1 of Maintenance cycle 3 and for the remaining duration of the study. Patients and their caregiver view the MIPE program that features video clips of ALL patients and their parents/other adults discussing Maintenance treatment in the clinic on day 1 of cycle 3. A designated parent/other adult is selected and trained briefly in prompting and supervising the patient to take 6MP daily by the CRA on day 1 of Maintenance cycle 3. Patients also receive customized printed medication schedules approximately every 4 weeks (days 1, 29, and 57) during Maintenance cycles 3-5 (during scheduled clinic visits) from their healthcare provider. Patients and/or the parent/other adult receive automated customized electronic reminders delivered via smartphone according to the patient's electronic 6MP schedule. Once the designated parent/other adult receives the reminder for 6MP, they are instructed to prompt initiation of the 6MP dose (if necessary), and to supervise the ingestion of the prescribed 6MP (in all instances). If the patient is not present when the dose of 6MP is due, the patient receives a call from the designated parent/other adult to prompt initiation of the dose. Patients and designated parents/other adults will be instructed to electronically indicate when 6MP has been taken (indicative of DST execution). If there is no response by the designated parent/other adult indicating 6MP ingestion within 1 hour of the scheduled time, additional automated reminders are sent. The Adherence Study Coordinating Center will evaluate electronic responses (indicative of DST execution) every 4 weeks. The DST response rates will be communicated to the COG sites, identifying the patients as low DST responders (response rate: < 85%) or high DST responders (response rate: ≥ 85%), along with instructions to serve as a guideline for communicating these results when reviewing them with their patient. DST response rates will be reviewed with the patient every 4 weeks at the clinic visit by the healthcare provider for all U-iIP patients (irrespective of response rate). Patients (and their designated caregiver) receive booster MIPE videos to view on their smartphone every 4 weeks (Days 1, 29, and 57) during Maintenance cycles 3-5, with content that reinforces the importance of 6MP in treating leukemia, having a daily routine for 6MP ingestion, and executing/confirming directly supervised therapy (DST) with each dose, and review common barriers to 6MP ingestion and DST execution (e.g., patient away from home, change in daily schedule), address additional barriers significantly associated with DST execution, and feature examples of patients/other adults self-identifying barriers (e.g., parent not always home at time of 6MP, lack of organizational skills, etc.), and provide specific steps to overcome the barriers. Additionally, patients undergo blood sample collection on the study.

ADHERERS: Patients are randomized to 1 of 2 arms during cycle 2 of Maintenance therapy.

ARM III (EDU: Patients receive another Patient Supply Kit and MEMS® TrackCap™ to use on day 1 of Maintenance cycle 3 and for the remaining duration of the study. Patients and their caregiver view the MIPE program that features video clips of ALL patients and their parents/other adults discussing Maintenance treatment in the clinic on day 1 of cycle 3. Additionally, patients undergo blood sample collection on the study.

ARM IV (pIP): Patients receive another Patient Supply Kit and MEMS® TrackCap™ to use on day 1 of Maintenance cycle 3 and for the remaining duration of the study. On day 1 of Maintenance cycle 3, patients and their caregiver view the MIPE program that features video clips of ALL patients and their parents/other adults discussing Maintenance treatment in the clinic. On day 1 of Maintenance cycle 3, the patient and a designated parent/other adult are trained to set daily reminders on their smartphones at the time the 6MP is due, and to use the "snooze" function to allow repeated reminders in case the medication cannot be taken when the alarm first goes off. The designated parent/other adult is also trained briefly by the CRA in prompting and supervising the patient to take 6MP daily. Once the designated parent/other adult hears the smartphone alarm for 6MP, they are instructed to prompt initiation of the 6MP dose (if necessary), and to supervise the ingestion of the prescribed 6MP (in all instances). If the patient is not present when the dose of 6MP is due, the patient receives a call from the designated parent/other adult to prompt initiation of the dose. Additionally, patients undergo blood sample collection on the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: >= 10 years and =< 25 years
* Previously enrolled onto AALL1732
* Consented to the AALL1732 mercaptopurine adherence correlative study
* Maintenance therapy has not yet begun
* English or Spanish-speaking (patient and parent/other adult)
* Planning to receive 6MP (as tablets) during maintenance phase of therapy
* Able and willing to use the MEMS® TrackCap™ (e.g., not using a pillbox or prescribed liquid 6MP)
* Has a designated parent/other adult who is willing to enter into a mutual agreement with the patient to participate in a daily supervised medication administration routine
* Patient/parent/other adult must be willing to use a smartphone to receive medication reminders
* Receiving treatment at a Children's Oncology Group (COG) institution in the United States

Exclusion Criteria:

* Patients who have previously participated in or are currently participating in another intervention clinical trial designed to improve adherence
* Regulatory requirements

  * All patients and/or their parents or legal guardians must sign a written informed consent
  * All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2027-03-03 (Estimated); Study Completion 2027-03-03 (Estimated)

PRIMARY OUTCOMES:
Participation | At baseline (by day 1 of maintenance chemotherapy)
  Will calculate and report the proportion of patients eligible for the study who participate and will report a corresponding 95% confidence interval.
Refusal reasons | At baseline (by day 1 of maintenance chemotherapy)
  A single question in a study case report form prompts refusal reason. For each available reason, will calculate and report the proportion of patients reporting that refusal reason as well as corresponding 95% confidence intervals.
Attrition | By 60 weeks from day 1 of maintenance chemotherapy
  Will calculate and report the proportion of patients who drop out of the study prior to completion among those eligible and enrolled and will report the corresponding 95% confidence interval.
Completion of study measures | By 60 weeks from day 1 of maintenance chemotherapy
  Will calculate and report the proportion of patients who complete the following measures by the end of the study follow-up period: study survey submission, MEMS® TrackCap™ return, maintenance form return, and blood sample submission. Will also report the corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
6-mercaptopurine (6MP) adherence (baseline non-adherers) | By 60 weeks from day 1 of maintenance chemotherapy
  Among baseline non-adherers, the proportion of days with protocol defined appropriate medication use during the study follow up period will be captured for each patient using the MEMS cap. Will calculate and report the mean proportion of adherence days by arm and the corresponding 95% confidence interval.
6MP adherence (baseline adherers) | By 60 weeks from day 1 of maintenance chemotherapy
  Among baseline adherers, protocol defined appropriate medication use during the study follow up period will be captured for each patient using the MEMS cap. Will calculate and report the proportion with >= 95% adherence over the study follow up period by arm with a corresponding 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Smita Bhatia, Principal Investigator — Children's Oncology Group
Locations (27):
- United States (27):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Oakland, Oakland, California
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Riley Hospital for Children, Indianapolis, Indiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin